CLINICAL TRIAL: NCT06401148
Title: Exercise-based Cardiac Rehabilitation for Patients with Atrial Fibrillation Receiving Catheter Ablation
Brief Title: Exercise-based Cardiac Rehabilitation for Atrial Fibrillation
Acronym: ExCR-AF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2024-04-19; First posted 2024-05-06 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise-based cardiac rehabilitation (Experimental): Participants will complete an 8-week-long cardiac rehabilitation programme consisting of supervised exercise sessions run by a clinical exercise physiologist and psychoeducation sessions.
  Interventions: Behavioral: Cardiac rehab intervention group
- Treatment as Usual (No Intervention): Participants randomised to usual care will not receive any intervention but continue with usual medical treatment for their AF as determined by their healthcare team.

INTERVENTIONS:
Behavioral: Cardiac rehab intervention group — Participants will complete an 8-week cardiac rehabilitation programme supported by the onsite CR service.
  Arms: Exercise-based cardiac rehabilitation

SUMMARY:
The investigators aim to conduct a pilot randomised controlled trial (RCT) with embedded feasibility study to evaluate an exercise-based cardiac rehabilitation (ExCR) programme when delivered to patients with atrial fibrillation on the waiting list for catheter ablation. Our overall objective is to test the feasibility and acceptability of an evidence-based ExCR intervention prior to evaluation in a future randomized controlled trial (RCT).

DETAILED DESCRIPTION:
A two-arm pilot randomised feasibility trial (RCT) with embedded process evaluation will be undertaken as a phased programme of work. Patients on a waiting list for catheter ablation will be offered a referral to cardiac rehabilitation. The intervention consists of supervised exercise sessions run by a clinical exercise physiologist and psychoeducation sessions. The trial will involve one National Health Service (NHS) research site, Liverpool Heart and Chest NHS Foundation Trust enrolling patients (n=60) to assess intervention and study design processes. Primary outcomes are recruitment rate, adherence to the ExCR and loss to follow-up. Semi-structured interviews and focus groups with patients and clinicians will be used to gather data on the acceptability of the intervention and study procedures. Secondary outcome measures will be taken at baseline (preintervention), postintervention and at 6 month follow-up for both phases and will consist of exercise capacity measured by AF burden, AF recurrence, quality of life, exercise capacity, and cardiac structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged ≥18 years.
* Diagnosed with AF and on a waiting list or referred for medical treatment for symptomatic AF (eg catheter ablation).
* Is eligible and willing to take part in an ExCR programme.

Exclusion Criteria:

* Blood pressure >180/100.
* Unstable angina.
* Severe valvular heart disease as diagnosed by echocardiography.
* Heart failure New York Heart Association (NYHA) class 4.
* <6 months post-transplant.
* Resting/uncontrolled tachycardia.
* Stroke in last 6 weeks.
* Cardiac sarcoidosis.
* Injury or disability preventing exercise.
* Inability to understand trial procedures e.g. difficulties with speaking and understanding the English language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients screened, eligible and approached | Baseline
  The percentage of patients that are screened, eligible and approached
  decline CR (including reasons for declining) agree to CR and consent to being part of the study The percentage of patients that take up standard CR and reasons for drop out; and the percentage of participants that complete outcome assessments and reasons for drop out.
Patient focus groups to assess intervention and testing acceptability | Up to 20 weeks from baseline
  Patient Focus Groups
Clinical exercise physiologist interview to assess intervention and testing acceptability | Up to 20 weeks from baseline
  Clinical Exercise Physiologist Interview

SECONDARY OUTCOMES:
Changes in AF burden | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  Changes in atrial fibrillation burden as measured by the University of Toronto Atrial Fibrillation Severity Scale (AFSS). The AFSS is a disease-specific measure used to capture subjective and objective ratings of disease burden in patients with atrial fibrillation. It assesses atrial fibrillation burden (score 1-30; higher scores indicate higher burden); Global Well Being (a visual analogue scale ranging from 1-10, indicating a patient reports as having a worst possible life [0] to the best possible life[10]); AF symptom score (score of 0-35; higher scores indicate more bothered by AF symptoms); and health care utilization (score of 0-21; higher scores indicate greater health care utilization).
AF Recurrence | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  AF recurrence will be measured using the AliveCor KardiaMobile which is a hand-held one lead electrocardiogram (ECG) device.
  Kardia Mobile is an FDA approved device that allows six lead ECG recording for 30 seconds using the patient's smart phone. The device has a automated algorithm that interprets the ECG as either 'sinus rhythm', 'AF', or 'unclassified'. We will be collecting the counts of these classifications to assess the number of AF episodes.
Disease specific quality of life measured by the AFEQT questionnaire | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  Health related quality of life as measured by the Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT). The AFEQT assesses 4 domains: symptoms, activities, treatment concern, treatment satisfaction, and a summary score that includes the first 3 domains. Patients will assess the impact of AF on their health status during the previous 4 weeks. Responses are presented on a 7-point Likert scale. Raw scores within each domain are transformed from a 0 (most severe symptoms) to a 100 scale (no limitations or disability).
General quality of life as measured by the EQ-5D-5L questionnaire | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  The 5-level EuroQol-5 Dimensions (EQ-5D-5L) is a parsimonious measure of health-related quality of life consisting of five dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. It also includes a Visual Analogue Scale (EQ-VAS) aimed at capturing participants' rating of their 'health today' on a scale from 0-100 with 100 being the best state and 0 being the worst state.
  The EQ-5D will also be used to inform economic evaluation.
VO2 peak measured via CPET | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  Maximal oxygen consumption (VO2peak) will be measured using cardiopulmonary exercise testing (CPET). Peak exhaustion will be evaluated by several variables (e.g. respiratory exchange ratio ≥T 1.10, heart rate and subjective exhaustion of the patient). VO2peak will be defined as the peak VO2 reached during the test. The test will be performed by two members of the research team. For safety reasons, pre-set criteria for initiation and/or termination of the test have been defined.
  Additional variables will include ventilatory thresholds (VT1 and VT2), VO2 slopes, and O2 pulse.
Exercise capacity measured via the 6MWT | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  The maximum walking distance (in metres) within 6 minutes will be used to assess exercise capacity, measured via the six-minute walk test (6MWT).
Cardiac structure and function measured via echocardiography | At baseline, post intervention (8-10 weeks) and 6 months after intervention
  Transthoracic Echocardiography (echo) will be performed by a clinically accredited echocardiographic. Cardiac structure and function will be assessed non-invasively with the participant lying on their left side. Standard 2-dimensional (2D), 3-dimensional (3D) Doppler, tissue-Doppler (TDI) and M Mode scans will be performed using a commercially available ultrasound system (Vivid iQ, GE Medical, Horton, Norway) with a 1.5-4 megahertz (MHz) phased array transducer applied to the participant's chest.
  A full level 2 transthoracic assessment in keeping with the British Society of Echocardiography) BSE minimum dataset, including left ventricular ejection fraction, left atrial volume, left atrial strain (and rate), left atrial volumetric function, left ventricle filling pressures, right atrial strain and exploratory 3D volumes.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Buckley, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fitzhugh C, Jones H, Foweather L, Lip GYH, Gupta D, Mills MT, Buckley BJ. Exercise-based cardiac rehabilitation for patients with atrial fibrillation receiving catheter ablation: protocol for a feasibility randomised controlled trial (RCT) with embedded process evaluation. BMJ Open. 2025 Jan 30;15(1):e088460. doi: 10.1136/bmjopen-2024-088460. PMID 39890138